CLINICAL TRIAL: NCT01766908
Title: Timing of Umbilical Cord Clamping After Vaginal or Cesarean Preterm Birth
Brief Title: Optimal Timing of Cord Clamping in Preterm Pregnancy Following Vaginal or Cesarean Delivery
Acronym: CordClamp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, James Martin, Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011-0270
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Preterm Birth
Keywords: Timing of Umbilical Cord clamping; Cord Clamp 20 seconds; Cord Clamp 40 seconds; Cord Clamp 60 seconds
MeSH Terms: conditions — Premature Birth | interventions — Cesarean Section

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cord Clamp 20 Seconds After Delivery (Active Comparator): Intervention is cord clamp at 20 seconds following vaginal or cesarean delivery
  Interventions: Other: Clamp cord 20, 40 or 60 seconds following vaginal or cesarean delivery
- Cord Clamp 40 seconds After Delivery (Active Comparator): Timing of cord clamp at 40 seconds following vaginal or cesarean delivery.
  Interventions: Other: Clamp cord 20, 40 or 60 seconds following vaginal or cesarean delivery
- Cord Clamp 60 seconds After Delivery (Active Comparator): Intervention is timing of cord clamp at 60 seconds following vaginal or cesarean delivery
  Interventions: Other: Clamp cord 20, 40 or 60 seconds following vaginal or cesarean delivery

INTERVENTIONS:
Other: Clamp cord 20, 40 or 60 seconds following vaginal or cesarean delivery — None to add
  Other Names: Clamping of umbilical cord following either preterm vaginal or cesarean delivery

SUMMARY:
This is an experimental research study for pregnant women between 23 and 37 weeks age of gestation who will be having a baby sooner than term. This study is to learn if waiting 20, 40, or 60 seconds to clamp the umbilical cord after baby delivers will improve his/her outcome and overall health. Benefit to the baby may come by increasing the amount of blood in the baby's body, reducing the need for possible transfusion later, and possible prevention of other complications caused by too little blood in the baby. Possible reduction of cerebral palsy may be realized by a longer interval for cord clamping.

DETAILED DESCRIPTION:
Intention is to enroll every preterm delivery into this trial containing six groups of patients, vaginal or cesarean delivery with clamping of the cord at 20, 40 or 60 seconds. Expectation is 1500 deliveries over 2 year period of time. Randomization upon entry to L&D unit. Removal from study if resuscitation deemed urgent by newborn staff. Strong effort to keep newborn warm using appropriate measures. Evaluation to determine if there are differences in transfusion, anemia, time to onset of spontaneous respiration, occurence of IVH or CP.

ELIGIBILITY:
Inclusion Criteria:

18 years old singleton gestation Between 23-37 weeks gestation Able to understand and sign informed consent

Exclusion Criteria:

multiple gestation/ known intrauterine fetal death unable to sign consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Intraventricular Hemorrhage number and severity | 15 months
  WE are seeking the length of time to delay cord clamping for various gestational age groups following vaginal or cesarean delivery in order to significantly improve primary outcome.

SECONDARY OUTCOMES:
Incidence and volume of red cell transfusion for newborns. | 15 months
  Benefits will be significantly better with very preterm deliveries compared to those delivered from 29-36 weeks gestation. These benefits will include a lower incidence of transfusion and less frequent/less severe intraventricular hemorrhage in new borns.

CONTACTS AND LOCATIONS:
Overall Officials: James Martin, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Winfred L. Wiser Hospital for Women and Infants, Jackson, Mississippi, United States